CLINICAL TRIAL: NCT05625750
Title: Study on the Characteristic, Therapy and Prognosis of Patients With Nonalcoholic Fatty Liver Disease
Brief Title: Observational Study About Patients Diagnosed With NAFLD
Status: Recruiting | Type: Observational
Sponsor: Xiangya Hospital of Central South University (Other)
Responsible Party: Principal Investigator, Huang Yan, Professor, Xiangya Hospital of Central South University
Other Study IDs: Xiangya NAFLD project
Record Dates: First submitted 2022-11-15; First posted 2022-11-23 (Actual); Last update posted 2022-11-30 (Actual); Status verified 2022-11

CONDITIONS: Nonalcoholic Fatty Liver Disease
Keywords: Nonalcoholic Fatty Liver Disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood including blood cells, serum and plasma, urine, faeces and liver tissue (if necessary)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients diagnosed with NAFLD: All subjects will receive the currently recognized routine test of NAFLD according to their disease and no additional intervention and treatment will be added for subjects

SUMMARY:
Nonalcoholic fatty liver disease (NAFLD) is the most common condition affecting the liver, owing to its association with obesity and the metabolic syndrome. The largest study to date using magnetic resonance spectroscopy to quantify liver triglyceride (TG) content showed that approximately 33% of individuals have hepatic steatosis. NAFLD encompasses a continuum of histological findings that starts with steatosis that can progress to nonalcoholic steatohepatitis (NASH), which is characterized by inflammation and cell death, and eventually cirrhosis. Given the large number of individuals afflicted with this condition, there is a clear need to develop effective and safe therapies to treat NAFLD.

DETAILED DESCRIPTION:
Patients with NAFLD were recruited in the current study and divided into NAFLD group, and NASH group. The researchers will collect various clinical examination indexes of the subjects in the process of diagnosis and treatment, including but not limited to ALT, AST, TG, TC, etc. Characteristic and prognosis of patients will be recorded. The serum, feces, urine and liver (if necessary) samples of all subjects will be taken after enrollment and stored for probably testing in the future. This study has no additional intervention and treatment for subjects.

ELIGIBILITY:
Inclusion Criteria:

1. patients diagnosed with nonalcoholic fatty liver disease

Exclusion Criteria:

1. patients suspected of excessive alcohol consumption
2. malignant tumors, dementia, active tuberculosis, AIDS, organ failure, pregnancy or breastfeeding, etc cannot cooperate with the investigation
3. incomplete data such as HBV serological results and abdominal ultrasound results
4. patients who refuse to sign informed consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients between the age of 18-75, who was diagnosed with NAFLD were all elligible for this observational study.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-04-27 (Actual); Primary Completion 2025-04-27 (Estimated); Study Completion 2027-04-27 (Estimated)

PRIMARY OUTCOMES:
BMI | 3 weeks
  BMI stands for body mass index. This is the ratio of a person's height to their weight.
alcohol intake | 3 years
  alcohol consumption every week

CONTACTS AND LOCATIONS:
Overall Officials: Yan Huang, Study Director — Xiangya Hospital of Central South University
Locations (1):
- Department of Infectious Disease, Xiangya Hospital, Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wang S, Zhu Q, Liang G, Franks T, Boucher M, Bence KK, Lu M, Castorena CM, Zhao S, Elmquist JK, Scherer PE, Horton JD. Cannabinoid receptor 1 signaling in hepatocytes and stellate cells does not contribute to NAFLD. J Clin Invest. 2021 Nov 15;131(22):e152242. doi: 10.1172/JCI152242. PMID 34499619